CLINICAL TRIAL: NCT05577039
Title: Preoperative Renal Resistive Index to Predict Long-term Development of Chronic Kidney Disease in Patients Undergoing Cardiac Surgery
Brief Title: Preoperative RRI and Long-term Risk for CKD
Status: Completed | Type: Observational
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Other Study IDs: K 2021-9906
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2022-10

CONDITIONS: Acute Kidney Injury; Acute Kidney Disease; Chronic Kidney Disease; Cardiac Surgery; Renal Resistive Index
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Renal resistive index (RRI) is calculated from ultrasonographic Doppler measurements of flow velocities in intraparenchymal renal arteries. Normal values are around 0.60, and 0.70 is considered the upper normal threshold in adults. Both preoperative and postoperative elevation of RRI has shown promise in early detection of AKI after cardiac surgery. Further, elevated RRI before coronary angiography is associated with an increased risk of cardiovascular complications up to 1 year after the procedure. The role of preoperative RRI in predicting long-term renal and cardiovascular complications after elective surgery is however not known. The aim of this study is to assess the role of preoperative RRI to predict the risk of persistent renal dysfunction as well as renal- and cardiovascular complications up to 5 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Elective coronary artery bypass grafting, heart valve surgery, or aortic surgery performed at Karolinska University Hospital between September 2014 and April 2015
* Preoperative measurement of RRI performed with satisfactory Doppler reading
* Written informed consent

Exclusion Criteria:

* Kidney transplant
* Dialysis-dependent kidney disease
* Cancelled surgery
* Missing follow-up data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective cardiac surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Long-term renal dysfunction | 5 years after surgery or end of follow-up
  Reduced estimated glomerular filtration rate (eGFR) ≥25% from baseline

SECONDARY OUTCOMES:
Short-term renal dysfunction | 30 days after surgery
  Reduced eGFR ≥25% from baseline
Intermediate renal dysfunction | 90 days after surgery
  Reduced eGFR ≥25% from baseline
Major adverse kidney events (MAKE) | 30 days, 90 days, 1 year, and 5 years after surgery or end of follow-up
  Composite outcome during follow-up time including one of; death, renal replacement therapy, reduced eGFR ≥25% from baseline
Major adverse cardiac and cerebrovascular events (MACCE) | 30 days, 90 days, 1 year, and 5 years after surgery or end of follow-up
  Composite outcome during follow-up time including one of; death, myocardial infarction, heart failure, stroke

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hertzberg, M.D., Principal Investigator — Department of Perioperative Medicine and Intensive Care, Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided